CLINICAL TRIAL: NCT05397353
Title: Sleep Treatment for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Old Dominion University (Other); Children's Hospital of The King's Daughters (Other)
Responsible Party: Principal Investigator, Evan M. Kleiman, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021001233
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sleep Problem; Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Parasomnias; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleepio (Experimental): Participants will receive the SleepioTM app
  Interventions: Other: Sleepio (TM)

INTERVENTIONS:
Other: Sleepio (TM) — Sleepio is a mobile Digital Cognitive Behavior Therapy for Insomnia (dCBT-I) app.

SUMMARY:
The purpose of this research study is to test a brief (6-session), empirically supported, and highly disseminable version of digital (i.e., smartphone or web-based) cognitive behavioral therapy for insomnia (dCBT-I), called SleepioTM, in suicidal adolescents with co-occurring insomnia during the high-risk post-hospitalization period. Suicide is the 2nd leading cause of death among adolescents. Sleep problems, such as insomnia symptoms-the most common sleep problem in youth-may be a particularly promising treatment target to reduce suicide risk in adolescents. The investigators propose to test the feasibility, acceptability, and effectiveness of dCBT-I in a two-site (Rutgers and Old Dominion University) pilot study trial. Adolescents, 14-18 years-old, recently hospitalized for suicide risk with co-occurring insomnia (n=20 pilot, 50% at each site), will receive dCBT-I (six weekly, 20-minute sessions) plus post-hospitalization treatment-as-usual (TAU). Adolescents will complete assessments pre-treatment, during the treatment phase including at the end of treatment, and 1-month follow-up post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18 years old (assessed via review of unit census).
* Recent psychiatric hospitalization due to suicide risk (i.e., suicide attempts, aborted/interrupted attempts, or suicide ideation with intent and/or a plan): assessed using an abbreviated version of the Columbia Suicide Severity Rating Scale (C-SSRS). In terms of recency, adolescents will need to enroll in the baseline assessment within three months of discharge from the hospital in order to assess the high-risk post-hospitalization period.
* Clinically significant insomnia symptoms: consistent with prior trials using the SleepioTM package, participants will be screened using the Sleep Condition Indicator (SCI)-an 8-item measure created by SleepioTM treatment developers to screen for DSM-5 insomnia disorder. The SCI assesses sleep duration, quality, and difficulties, and daytime impairment due to sleep problems; lower scores on the SCI indicate poorer sleep conditions and a cutoff of ≤16 indicates probable insomnia disorder, which will be the cutoff used for the current study.
* Motivation to engage in sleep treatment: consistent with other trials testing SleepioTM, questions will be used to assess perception of sleep problem severity and desire to change. The scale includes (1) "At present, sleep is a big problem for me" and (2) "I want to change my sleep" rated on a scale 0=strongly disagree to 10=strongly agree. Each item must be rated ≥5, in line with prior trials. Given this is a digital intervention, this criterion will help ensure we recruit adolescents who are likely to engage with treatment. Importantly, we note that prior trials have not needed to exclude anyone based on this criterion, reflecting the idea that the majority of participants we encounter will be motivated to engage in this novel treatment.

Exclusion Criteria:

Prior CBT-I treatment (the intervention being tested in this study): prior treatment would indicate non-response to a reasonable dose of this empirically supported treatment.

* At high risk for obstructive sleep apnea (OSA): The STOP-BANG sleep apnea screening questionnaire (modified for adolescents) will be used to screen adolescents at high risk for OSA, who will be referred for a non-study polysomnography screening.
* Bipolar disorder: given concerns that certain components of CBT-I (i.e., sleep restriction) may be risky for this population.
* Substance use disorder that is primary to insomnia: significant substance use (alcohol or drug) disorders would require alternative treatment.
* Presence of factors that may reduce participant's ability to provide assent/consent or to complete the study procedures (e.g., non-English speaking, severe cognitive impairment, pervasive developmental disorder, acute psychosis, risk for other-directed violence).
* Unwillingness to wear the actigraphy device or to complete smartphone-based EMA at the time of enrollment: consistent with the research team's prior studies, if participants are actively enrolled in the study and then decide that they no longer want to wear the wrist actigraphy device, we will give them the option to continue only the SleepioTM and smartphone-based EMA parts of the study. • Not having a parent/legal guardian willing to provide permission (if adolescent is a minor) or consent (for their own participation): although permission is only required for minors, parents will be included for all adolescents to keep study procedures consistent for all participants.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | up to 10 weeks
  Insomnia Severity Index (same measure as baseline) assessed weekly from the beginning of treatment until the treatment is complete (or a maximum of 10 weeks to match assessment with the TAU only group).
Suicidal thoughts | up to 10 weeks
  Suicide ideation severity will be measured weekly with the Beck Suicide Ideation Scale (same measure as baseline) until the end of treatment.

SECONDARY OUTCOMES:
Sleep problems | daily through study completion, up to 10 weeks
  The following sleep parameters will be assessed using a combination of daily sleep diaries (EMA app) and wrist actigraphy (Actiwatch). (a) sleep efficiency (SE): % of time in bed spent asleep; (b) sleep onset latency (SOL): how many minutes it takes to fall asleep; (c) total sleep time (TST): actual time slept (out of time in bed); (d) wake after sleep onset (WASO): total amount of time awake during the night; and (e) sleep quality: subjective ratings on 1=very poor to 5=very good.
Daily Suicidal Thoughts | daily through study completion, up to 10 weeks
  Daily reports of suicide ideation from EMA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rutgers University Behavioral Healthcare, Piscataway, New Jersey
  - Old Dominion University, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in accordance with NIMH Data Archive Agreement
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after the study is complete
Access Criteria: Registration on NIMH Data Archive

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT05397353/ICF_000.pdf